CLINICAL TRIAL: NCT00592020
Title: "Short Transverse" Versus Conventional "Hockey Stick" Incision in Kidney Transplantation
Brief Title: Short Transverse Versus Conventional Hockey Stick Incision in Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Daniel Inderbitzin, Clinic of Visceral and Transplant Surgery, University Hospital Inselspital, Bern
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 220/07
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Kidney Transplantation
Keywords: kidney; transplantation; minimal invasive; short transverse; hockey stick; incision; quality of life; planned kidney transplantation
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Short Transverse Incision
  Interventions: Procedure: Short Transverse Incision
- 2 (Active Comparator): Hockey Stick Incision
  Interventions: Procedure: Hockey Stick Incision

INTERVENTIONS:
Procedure: Short Transverse Incision — Short Transverse Incision for kidney transplantation
  Arms: 1
Procedure: Hockey Stick Incision — Hockey Stick Incision for kidney transplantation
  Arms: 2

SUMMARY:
Today the minimal invasive access is used for a lot of different operations. This technique takes the advantage of less postoperative pain, better cosmetic results, and a lower surgical complication rate (e.g. hernia, wound infection).

Especially patients under immunosuppressive therapy could benefit from this technique. First results in minimally invasive kidney transplantation indicate that it may be performed quickly and safely. Benefits are expectable on postoperative pain, recovery, and surgical complications. Another retrospective study showed lower rates of hernia, abdominal wall relaxations, and a better postoperative cosmetic.

The aim of this study is to compare the classic hockey stick incision with a minimal invasive incision in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or over 18 years
* Sole kidney transplantation
* Consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
QoR (Quality of Recovery) - Score | preoperative, day 1/3/5/7 postoperative

SECONDARY OUTCOMES:
Quality of Life by SF (Short Form) 36 | preoperative, day 7, week 4, month 6 postoperative
Operation time | intraoperative
Warm ischemic time | intraoperative
Postoperative pain measured by VAS (visual analog scale) and amount of analgesia | day 1/2/3/4/5/6/7 postoperative
Surgical complications | day 7, week 4, month 6, month 12 postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Uta Herden, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Inselspital, Bern, Canton of Bern, Switzerland